CLINICAL TRIAL: NCT05177653
Title: Separate and Combined Extrapancreatic Effects of Glucose-dependent Insulinotropic Polypeptide and Glucagon-like Peptide 1
Brief Title: Separate and Combined Extrapancreatic Effects of the Incretin Hormones
Acronym: GA-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-21035117
Record Dates: First submitted 2021-11-16; First posted 2022-01-04 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pancreatectomy; Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — Infusions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GIPRA (Experimental)
  Interventions: Other: Intravenous infusion
- GLP-1RA (Experimental)
  Interventions: Other: Intravenous infusion
- GIPRA + GLP-1RA (Experimental)
  Interventions: Other: Intravenous infusion
- Saline (Placebo Comparator)
  Interventions: Other: Intravenous infusion

INTERVENTIONS:
Other: Intravenous infusion — GIP receptor antagonist (GIP(3-30)NH2)
  Arms: GIPRA
Other: Intravenous infusion — GLP-1 receptor antagonist (exendin(9-39)NH2)
  Arms: GLP-1RA
Other: Intravenous infusion — GIP(3-30)NH2 and exendin(9-39)NH2
  Arms: GIPRA + GLP-1RA
Other: Intravenous infusion — Saline
  Arms: Saline

SUMMARY:
The two gut-derived hormones, glucose-dependent insulinotropic polypeptide (GIP) and glucagon-like peptide 1 (GLP-1) is secreted from intestinal cells in relation to a meal and increase insulin secretion from the pancreas. The hormones also exert effects outside the pancreas, but especially for GIP, these are poorly investigated. Because of this, only GLP-1 based drugs (GLP-1 receptor agonists) are on the market for the treatment of type 2 diabetes and obesity. Nonetheless, a new drug is in clinical development: a combined GIP-GLP-1-receptor agonist (tirzepatide), which has shown better results than GLP-1 alone. The mechanism behind these impressive effects are unknown and in this study, the investigators will look into the exptrapancreatic effects of GIP and GLP-1, separate and combined and thus elucidate the mechanisms of action of this new drug class.

ELIGIBILITY:
Inclusion Criteria:

* Total pancreatectomy
* Caucasians
* Blood haemoglobin >7 mmol/l for males and >6.5 mmol/l for females

Exclusion Criteria:

* Pancreatectomy within the last 3 months
* Ongoing chemotherapy or chemotherapy within the last 3 months
* Treatment with GLP-1R agonists within the last 3 months
* Renal impairment (estimated by eGFR <60 ml/min/1.73 m2) and/or albuminuria
* Calcium related disease, hypo-/hyperthyroidism
* Known significant liver disease, ALT or AST >3 times normal value or INR outside normal range
* Severe arteriosclerotic heart disease or heart failure (NYHA group III or IV)
* Pregnancy and/or breastfeeding
* Use of more than 14 units of alcohol per week or abuse of narcotics
* Any condition that the investigator feels would interfere with trial participation

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Changes in plasma levels of glucose between interventions assessed through frequently blood sampling during the experimental days | Up to two months
  mmol/l
Changes in plasma levels of glucagon (gut-derived) between interventions assessed through frequently blood sampling during the experimental days | Up to two months
  pmol/l
Changes in plasma levels of insulin/C-peptide between interventions assessed through frequently blood sampling during the experimental days | Up to two months
  pmol/l
Changes in plasma triglycerides between interventions assessed through frequently blood sampling during the experimental days. | Up to two months
  mmol/l lipoproteins, neutral and complex lipids.
Changes in plasma lipoproteins between interventions assessed through frequently blood sampling during the experimental days. | Up to two months
  mg/dl
Changes in brown adipose tissue activity between interventions, assessed by thermographic camera | Up to two months
Changes in adiponectin in plasma between interventions, assessed through frequently blood sampling during the experimental days. | Up to two months
  μg/mL
Changes in CTX between interventions assessed through frequently blood sampling during the experimental days | Up to two months
  ng/ml
Changes in plasma P1NP between interventions assessed through frequently blood sampling during the experimental days | Up to two months
  ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Clinical Metabolic Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No